CLINICAL TRIAL: NCT05333276
Title: A Phase I Study of the TQB3602 Capsule Combined With AK105 Injection in Patients With Advanced Cancers
Brief Title: Clinical Trial of the TQB3602 Capsule Combined With AK105 Injection in Patients With Advanced Cancers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3602-AK105-I-01
Record Dates: First submitted 2022-04-12; First posted 2022-04-18 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Advanced Cancers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3602 Capsule + AK105 Injection (Experimental): TQB3602 capsule administered orally on day 1, 8 in 21-day cycle; every three weeks intravenous (IV) for one times of AK105 injection.
  Interventions: Drug: TQB3602 Capsule + AK105 Injection

INTERVENTIONS:
Drug: TQB3602 Capsule + AK105 Injection — TQB3602 is a kind of proteasome inhibitor, AK105 is an anti-PD-1 antibody.

SUMMARY:
TQB3602 is a kind of proteasome inhibitor, AK105 is an anti-programmed cell death protein 1 (PD-1) antibody.

ELIGIBILITY:
Inclusion Criteria:

* 1 Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
* 2 Age ≥ 18; Eastern Cooperative Oncology Group perfomance status score: 0-2; at least 3 months expected survival period.
* 3 Subjects with relapse advanced malignant solid tumors clearly diagnosed by pathology and / or cytology, lack of conventional effective treatment methods, failure or relapse after treatment.
* 4 Resolved acute effects of any prior therapy to baseline severity or Grade ≤ 1 per CTCAE v5.0 except for AEs not constituting a safety risk by investigator judgment.
* 5 Must have adequate organ and bone marrow function.
* 6 Male and female patients of childbearing potential and at risk for pregnancy must agree to use two highly effective method(s) of contraception throughout the study and for at least 6 months after the last dose of assigned treatment.

Exclusion Criteria:

* 1 Subjects with other malignancies currently or suffered within 3 years. The following two conditions can be enrolled: other malignant tumors treated with a single operation to achieve disease-free survival (DFS) for 5 consecutive years; cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors[ Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
* 2 Sujects with multiple factors affecting oral administration；
* 3 Subjets with unhealed toxicity above Grade 1 Common Terminology Criteria for Adverse Events Version 5.0 due to previous antitumor treatment；
* 4 Subjects who have received major surgical treatment, open biopsy or obvious traumatic injury within 4 weeks before first administration；
* 5 Subjects who have received surgery, chemotherapy, radiotherapy or other anticancer therapies 4 weeks before the first administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | During the first 21 days
  DLT will be assessed during the first 21 days of treatment for dose-escalation and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (21 days) of treatment.
Maximum tolerated dose (MTD) | During the first 21 days
  MTD is defined as the highest dosing schedule cohort level at which no more than 1 of 6 patients experience a Dose Limiting Toxicity (DLT).
Recommended phase II dose (RP2D) | Up to Cycle 28 (Cycle Length= 21 days)
  The RP2D was the maximum tolerated dose (MTD) or less.

SECONDARY OUTCOMES:
Number of patients with adverse events (AEs) and serious adverse events (SAEs) | From the time of informed consent signed to 90 days after the last dose
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Progression-free survival (PFS) | up to 2 years
  Defined as the time from the first dose of TQB3602 and AK105 to the first occurrence of disease progression or death from any cause.
Disease control rate (DCR) | up to 2 years
  Defined as the proportion of subjects with CR (Complete response), PR (Partial response), or SD (Stable Disease).
Duration of Response (DOR) | up to 2 years
  Defined as the time from first documented response to documented disease progression.
Overall survival (OS) | up to 5 years
  OS is defined as the time between the date of first administration and the date of death due to any cause. A participant who has not died will be censored at the last known alive date.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Nong Yang, Changsha, Hunan